CLINICAL TRIAL: NCT03029130
Title: Does Extending Catheterization Improve Outcomes in Early Vesicovaginal Fistula Repair Failures? A Prospective Randomized Controlled Trial
Brief Title: Catheter Extension Trial for Early Vesicovaginal Fistula Repair Failures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Evangel VVF Centre (Other)
Responsible Party: Principal Investigator, Steven Shephard, Fistula Surgeon, Evangel VVF Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EvangelWFC
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Vesico Vaginal Fistula
Keywords: vesicovaginal fistula; urinary catheter; catheter extension
MeSH Terms: conditions — Vesicovaginal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter Extension (Experimental): Patients in this arm will have a foley catheter re-passed, to remain in situ for an additional 14 days, after which time the catheter will be removed and the patient discharged to return for follow up exam at 3 months postop.
  Interventions: Device: Catheter extension
- Discharge (No Intervention): Patients in this arm will be discharged, to return for follow up exam at 3 months postop.

INTERVENTIONS:
Device: Catheter extension — Foley transurethral catheter placed to allow continuous drainage of urine.
  Arms: Catheter Extension

SUMMARY:
This study evaluates the use of extending time of continual urinary drainage (using transurethral foley catheter) for patients with early failures of vesicovaginal fistula repairs. Half of those included will be randomized to replacement of foley catheter for a length of 14 additional days, while the other half will be discharged (no intervention). Both groups will be examined for outcomes at 3 months post-repair.

DETAILED DESCRIPTION:
At present, there is no standard of care nor consensus for the proper management of repaired vesicovaginal fistulas that begin leaking prior to or immediately after scheduled catheter removal. In the past, extension of time with catheterization has been tried, with patients becoming fully healed by the time of catheter removal. However, some patients who are discharged with a fistulous leak later return at follow up completely dry, with a closed and healed fistula. This study will compare, in a prospective, randomized manner, extension of catheterization vs no intervention, to see if in such patients extending catheterization will improve their likelihood of complete fistula healing.

ELIGIBILITY:
Inclusion Criteria:

* Women who present with a vesicovaginal fistula for surgical repair AND who, at the time of initial catheter removal (7 or 14 days post-repair), have demonstrable fistulous leak on dye test

Exclusion Criteria:

* HIV infection,
* concomitant bladder stone(s),
* one or more ureters outside of the bladder,
* urethrovaginal fistula,
* multiple fistulas (more than one),
* dye leak / fistulous leak present at end of surgical procedure,
* radiation-induced fistula,
* fistula caused by cancer or infection (such as lymphogranuloma venereum),
* continence procedures being performed (such as pubovaginal sling),
* rectovaginal fistula,
* pregnancy,
* fistula breakdown of greater than 2cm identified on postoperative dye test.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Fistula closure | 3 months post-repair
  Successful closure of the fistula, as defined by patient self-reporting no urinary leakage AND a negative dye test proving no fistulous leak

SECONDARY OUTCOMES:
Urinary continence | 3 months post-repair
  Patient is completely continent of urine with no reported OR demonstrable leakage of dye on inspection.
Closure and continence at hospital discharge | Date of discharge (7-28 days post-repair)
  Rates of fistula closure and complete urinary continence at the time of hospital discharge
Complications | Duration of hospitalization (minimum 7 days, maximum 28 days post-repair)
  Rates of complications or urinary tract infections during hospitalization

IPD SHARING:
Plan to Share IPD: No